CLINICAL TRIAL: NCT07064694
Title: Hybrid Parastomal Endoscopic Repair (HyPER): Ten-Year Experience and Lessons Learned From a Single-Center Cohort of 200 Patients
Brief Title: HyPER - Hybrid Parastomal Endoscopic Repair
Acronym: HyPER
Status: Completed | Type: Observational
Sponsor: Swissmed Hospital (Other)
Collaborators: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Other Study IDs: HyPER-200
Record Dates: First submitted 2025-07-05; First posted 2025-07-15 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Parastomal Hernia
Keywords: HyPER; parastomal hernia; abdominal wall surgery; Hernioplasty; Hernia
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HyPER Procedure: Combined laparoscopic and open surgical technique for parastomal hernia repair, including adhesiolysis, sac excision, mesh implantation, and stoma relocation if needed.
  Interventions: Procedure: Hybrid Parastomal Endoscopic Repair (HyPER)

INTERVENTIONS:
Procedure: Hybrid Parastomal Endoscopic Repair (HyPER) — Combined laparoscopic and open surgical approach involving adhesiolysis, hernia sac excision, intraperitoneal mesh fixation, and stoma revision or relocation as indicated. Standard mesh used was DynaMesh-IPST®; in selected cases, a cost-effective modification with macroporous polypropylene mesh and omental interposition was applied.

SUMMARY:
Retrospective single-center study analyzing long-term outcomes of Hybrid Parastomal Endoscopic Repair (HyPER) in 200 patients with symptomatic parastomal hernias, including recurrence, complications, and quality of life.

DETAILED DESCRIPTION:
This is a retrospective, single-center observational study evaluating surgical management of symptomatic parastomal hernias using a standardized Hybrid Parastomal Endoscopic Repair (HyPER) technique. The HyPER method integrates laparoscopic and open approaches to enable comprehensive dissection, mesh reinforcement, and anatomical correction, including stoma relocation and soft tissue reconstruction when indicated.

All patients were classified preoperatively according to the European Hernia Society (EHS) classification. The procedure included laparoscopic adhesiolysis, open excision of the hernia sac, and laparoscopic intraperitoneal mesh fixation. A synthetic mesh (typically DynaMesh-IPST®) was used in most cases. In selected patients, a cost-effective alternative mesh was applied using a technique referred to as the "Baldachin modification," with an omental flap interposed to prevent adhesions.

The study included adult patients with symptomatic parastomal hernias who underwent elective surgery at a tertiary referral center for abdominal wall reconstruction. Exclusion criteria involved disseminated malignancy, contraindications to laparoscopy, and severely limited life expectancy. Patients were followed up in a dedicated outpatient setting with regular clinical and imaging assessments.

The aim of this study was to evaluate feasibility, safety, and the potential for broad implementation of the HyPER technique in the surgical treatment of parastomal hernias.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Symptomatic parastomal hernia requiring surgical intervention
* Eligibility for elective surgery
* Preoperative classification using the European Hernia Society (EHS) system

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Disseminated malignancy
  * Contraindications to laparoscopy
  * Severely limited life expectancy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2024-08 (Actual); Study Completion 2024-08 (Actual)

PRIMARY OUTCOMES:
Recurrence rate of parastomal hernia | Up to 10 years postoperatively (mean follow-up 61 months)
  Proportion of patients with clinically or radiologically confirmed recurrence of parastomal hernia following the HyPER procedure, as assessed during routine follow-up.

SECONDARY OUTCOMES:
Postoperative complications | Within 30 days postoperatively
  Incidence of postoperative complications such as wound infections, seromas, bowel injury, and stoma-related issues requiring medical or surgical management.
Patient-reported quality of life | Baseline and last follow-up (up to 10 years)
  Patient-reported outcomes assessed using the Visual Analog Scale for Quality of Life (VAS-QoL), a 10-point scale ranging from 0 (worst possible health state) to 10 (best possible health state). Higher scores indicate improved physical comfort and psychosocial well-being. Preoperative and postoperative scores were collected during follow-up visits and compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Bielański Hospital, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in this study (including text, tables, and figures) will be made available upon reasonable request to qualified researchers whose proposed use of the data has been approved by the study team and the institutional ethics board. Data will be shared for the purpose of academic, non-commercial research only. Interested investigators should contact the corresponding author by email.
Time Frame: Beginning 6 months after publication; available for 5 years.
Access Criteria: Access will be granted following review and approval of a research proposal and execution of a data use agreement.

REFERENCES:
- [Background] Szczepkowski M, Zamkowski M, Alicja S, Piotr W, Smietanski M. Evaluating EHS parastomal hernia classification for surgical planning: a retrospective analysis of 160 consecutive cases in a single center. Hernia. 2024 Oct;28(5):1915-1923. doi: 10.1007/s10029-024-03121-w. Epub 2024 Aug 10. PMID 39123085
- [Background] Szczepkowski M, Przywozka-Suwala A, Ziolkowski B, Witkowski P, Perea J. Hybrid parastomal hernia endoscopic repair (HyPER): novel approach to parastomal hernia surgery. Br J Surg. 2024 Apr 3;111(4):znae092. doi: 10.1093/bjs/znae092. No abstract available. PMID 38593041
- [Background] Szczepkowski M, Skoneczny P, Przywozka A, Czyzewski P, Bury K. New minimally invasive technique of parastomal hernia repair - methods and review. Wideochir Inne Tech Maloinwazyjne. 2015 Apr;10(1):1-7. doi: 10.5114/wiitm.2015.50052. Epub 2015 Apr 14. PMID 25960785
- [Background] Smietanski M, Szczepkowski M, Alexandre JA, Berger D, Bury K, Conze J, Hansson B, Janes A, Miserez M, Mandala V, Montgomery A, Morales Conde S, Muysoms F. European Hernia Society classification of parastomal hernias. Hernia. 2014 Feb;18(1):1-6. doi: 10.1007/s10029-013-1162-z. Epub 2013 Oct 1. PMID 24081460
- [Background] Antoniou SA, Agresta F, Garcia Alamino JM, Berger D, Berrevoet F, Brandsma HT, Bury K, Conze J, Cuccurullo D, Dietz UA, Fortelny RH, Frei-Lanter C, Hansson B, Helgstrand F, Hotouras A, Janes A, Kroese LF, Lambrecht JR, Kyle-Leinhase I, Lopez-Cano M, Maggiori L, Mandala V, Miserez M, Montgomery A, Morales-Conde S, Prudhomme M, Rautio T, Smart N, Smietanski M, Szczepkowski M, Stabilini C, Muysoms FE. European Hernia Society guidelines on prevention and treatment of parastomal hernias. Hernia. 2018 Feb;22(1):183-198. doi: 10.1007/s10029-017-1697-5. Epub 2017 Nov 13. PMID 29134456